CLINICAL TRIAL: NCT03599908
Title: Evaluation and Validation of Novel Diagnostic Tool for Allergists (AbioSCOPE) in Volunteer Population With Respiratory Allergies
Brief Title: Evaluation and Validation of Novel Diagnostic Tool for Allergists (AbioSCOPE)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Abionic SA (Industry)
Responsible Party: Principal Investigator, François Spertini, Professor/Doctor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 309/12
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Allergic Rhinitis; Asthma
Keywords: IgE; skin prick tests; diagnosis; rhinitis; asthma; allergy; laboratory
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Disease; Rhinitis; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Venous blood collection prepared to obtain serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, investigators evaluated for the first time the diagnostic efficacy of abioSCOPE® versus Phadia Laboratory System as an aid in the diagnosis of allergic diseases. Investigators targetted the agreement between test results obtained in abioSCOPE® and a laboratory reference method (Phadia Laboratory System, ThermoFisher Scientific, Uppsala, Sweden), considered as a quasi-gold standard in IgE (immunoglobulin E) antibody assays. Investigators also reported the medical decision taken by a panel of allergy experts who had access to patient history, skin tests and IgE antibody assay, but blinded to the method used, i,e, the reference method or the abioSCOPE® .

ELIGIBILITY:
Inclusion Criteria:

* Subjects examined at ambulatory medicine medicine center CHUV / PMU and for wich serum sample is required for the research of specific IgE (allergic patients, allergic group) or for any other reason (immunological) (non-allergic control patients, control group)
* Subjects for which it is expected (allergic group subjects) or who will be asked (non-allergic control group) to perform a panel of standard prick tests as basic allergological investigation, including pollen birch, grasses, mites (D pter, D far), cat dander.
* Obtain informed consent from each subject before any study procedure.

Exclusion Criteria:

* Presence of positive HIV-1 viremia by the ultra-sensitive method in the 12 months preceding the study.
* Use of any investigational or non-registered product (drug or vaccine)
* Chronic administration (more than 14 days) of immunosuppressive or immunomodulatory drugs in the 6 months preceding the study for corticosteroids. This means a dose of Prednisone or equivalent substance greater than or equal to 0.5 mg per kg / day. Inhaled topical steroids are allowed.
* Administration of any immunoglobulin, any immunotherapy or administration of some blood products in the 3 months preceding the study, or planned during the study period.
* Any health condition or patient history, in the opinion of the investigator, could interfere with the evaluation of the study's objectives.
* Participation in another experimental protocol during the period of the study.
* Demonstration, confirmation or suspicion of a condition of immunosuppression or immunodeficiency (including HIV infection) based on medical history and physical examination (no laboratory test).
* A family history of congenital or hereditary immunodeficiency.
* Subjects taking any of the following medications: antihistamines in the week preceding the consultation, systemic steroids (inhaled or nasal steroids are allowed), anti-cytokines or cytokines, systemic interferon (injection local interferon α for the treatment of HPV is allowed) or treated with systemic chemotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with history of allergic rhinitis and asthma
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Diagnostic agreement between AbioSCOPE and Phadia Laboratory System | 12 months
  Comparison of the diagnostic agreement obtain went clinical samples are measured with AbioSCOPE or with Phadia Laboratory System

CONTACTS AND LOCATIONS:
Overall Officials: Francois Spertini, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois